CLINICAL TRIAL: NCT03262324
Title: Reliability and Validity of the Turkish Version of the Visual Analogue Scale Foot and Ankle (VAS-FA)
Brief Title: The Aim of Study is Translate and Adapt the Visual Analog Scale Foot and Ankle (VAS-FA) Instrument Into Turkish and Psycho-metrically Test Its Reliability and Validity Among Patients Who Had Foot and Ankle Disorders or Surgery
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant Professor of Physiotherapy and Rehabilitation, Hasan Kalyoncu University
Other Study IDs: 2017-09
Record Dates: First submitted 2017-08-24; First posted 2017-08-25 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ankle Injuries and Disorders; Foot Injuries and Disorders
Keywords: Foot and Ankle; Disorders; Outcome Measure
MeSH Terms: conditions — Ankle Injuries; Disease; Foot Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VAS-FA Turkish version — Self-reported outcome questionnaires
  Other Names: Foot Function Index; Short Form-36

SUMMARY:
There have previously been no validated a specific foot and ankle patient-reported outcome measures in Turkish. The Visual Analogue Scale Foot and Ankle (VAS-FA) will translated and adapted into Turkish language. Thereafter, 200 patients who had foot and ankle disorders or surgery will complete VAS-FA questionnaire set on two separate occasions. Analyses included testing of ﬂoor-ceiling effect, internal consistency, reproducibility, and validity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Participants who have foot and ankle disorders
* Participants must have an orthopedic intervention last 3 months;

  1. Conservative intervention
  2. Surgery intervention

Exclusion Criteria:

* Age less than 18 or more than 65
* Positive medical history concerning the entire lower extremity,

  1. Diabetes mellitus
  2. Drug abuse
  3. Psychiatric diseases
  4. Rheumatoid arthritis
  5. Neurological diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants must be sedentary person from Turkey and receiving treatment intervention between study dates for ankle or foot disorders
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
VAS-FA Turkish version | 1 week
  The VAS-FA contains 20 questions for the patient with ﬁve possible answers. For each question a VAS-value from 0 to 100 points is possible. The total value for the entire score (all 20 questions answered) is therefore 0-2000 points. This total value is then divided by 20, resulting in a possible total score ranging from 0 to 100 points.

SECONDARY OUTCOMES:
Foot Function Index (FFI) | 1 week
  It is a self-administered index consisting of 23 items divided into three subscales. To obtain a subscale score, the item scores for subscales are totaled and then divided by the maximum total possible for all of the subscale items that the patient indicates is applicable. Therefore, subscale scores range from 0 to 100, with higher scores indicating greater impairment. A total foot function score is derived by calculating the average of the three subscale scores.
Short Form-36 (SF-36) | 1 week
  Completion of the 36 items yielded an 8-subscale profile of patient functional health and well being, as well as empirically derived physical and mental health component summary (PCS and MCS) measures. The subscales are scored as percentages and the summary measures are scaled to provide a score out of 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, PhD, Study Director — Hasan Kalyoncu University; Günseli Usgu, Phd, Principal Investigator — Hasan Kalyoncu University; Can Muslu, MD, Study Chair — İstanbul Haseki Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Hasan kalyoncu üniversity, Gaziantep
  - İstanbul Haseki Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hunt KJ, Hurwit D. Use of patient-reported outcome measures in foot and ankle research. J Bone Joint Surg Am. 2013 Aug 21;95(16):e118(1-9). doi: 10.2106/JBJS.L.01476. PMID 23965711
- [Result] Angthong C, Chernchujit B, Suntharapa T, Harnroongroj T. Visual analogue scale foot and ankle: validity and reliability of Thai version of the new outcome score in subjective form. J Med Assoc Thai. 2011 Aug;94(8):952-7. PMID 21863677
- [Result] Richter, M., Zech, S., Geerling, J., Frink, M., Knobloch, K., & Krettek, C. (2006). A new foot and ankle outcome score: Questionnaire based, subjective, Visual-Analogue-Scale, validated and computerized. Foot and ankle surgery, 12(4), 191-199.
- [Result] Nair AV, Shamsuddin K, John PS, Hamalainen JA, Kurien MA. Correlation of visual analogue scale foot and ankle (VAS-FA) to AOFAS score in malleolar fractures using Indian language questionnare. Foot Ankle Surg. 2015 Jun;21(2):125-31. doi: 10.1016/j.fas.2014.10.006. Epub 2014 Dec 12. PMID 25937413
- [Result] Stuber J, Zech S, Bay R, Qazzaz A, Richter M. Normative data of the Visual Analogue Scale Foot and Ankle (VAS FA) for pathological conditions. Foot Ankle Surg. 2011 Sep;17(3):166-72. doi: 10.1016/j.fas.2010.05.005. Epub 2010 Jun 2. PMID 21783078
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Lin CW, Moseley AM, Refshauge KM, Bundy AC. The lower extremity functional scale has good clinimetric properties in people with ankle fracture. Phys Ther. 2009 Jun;89(6):580-8. doi: 10.2522/ptj.20080290. Epub 2009 May 7. PMID 19423644
- [Result] Button G, Pinney S. A meta-analysis of outcome rating scales in foot and ankle surgery: is there a valid, reliable, and responsive system? Foot Ankle Int. 2004 Aug;25(8):521-5. doi: 10.1177/107110070402500802. PMID 15363371
- [Result] Goldstein CL, Schemitsch E, Bhandari M, Mathew G, Petrisor BA. Comparison of different outcome instruments following foot and ankle trauma. Foot Ankle Int. 2010 Dec;31(12):1075-80. doi: 10.3113/FAI.2010.1075. PMID 21189208
- [Result] Repo JP, Tukiainen EJ, Roine RP, Kautiainen H, Lindahl J, Ilves O, Jarvenpaa S, Hakkinen A. Reliability and validity of the Finnish version of the Visual Analogue Scale Foot and Ankle (VAS-FA). Foot Ankle Surg. 2018 Dec;24(6):474-480. doi: 10.1016/j.fas.2017.05.009. Epub 2017 Jun 7. PMID 29409192